CLINICAL TRIAL: NCT02505815
Title: Neurocognitive Function After Regional and General Anesthesia: a Randomized Control Trial
Brief Title: Neurocognitive Function After Regional and General Anesthesia (245_14 B)
Acronym: 245_14_B
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2015-06-11; First posted 2015-07-22 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Neurocognitive Function
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Regional Anesthesia: Patients with surgery in regional anesthesia.
  Interventions: Procedure: Surgery; Procedure: Cortisol Level Measurement; Procedure: Neurocognitive Testing
- General Anesthesia: Patients with surgery in general anesthesia.
  Interventions: Procedure: Surgery; Procedure: Cortisol Level Measurement; Procedure: Neurocognitive Testing

INTERVENTIONS:
Procedure: Surgery
Procedure: Cortisol Level Measurement
Procedure: Neurocognitive Testing

SUMMARY:
Postoperative cognitive dysfunction (POCD) is a disease with restricted cognitive memory function and intellectual skills, which occurs after surgery with and without anesthesia. The POCD strongly depends on patient's age and the surgical operation type. The anesthesia procedure plays a pivotal role as well and regarding the current knowledge it is still uncertain which technique matches the lowest risk. Elevated stress level accompanied with regional anesthesia procedures are accused to cause POCD in elderly patients. The investigators address the question weather regional or general anesthesia leads to a pronounced POCD in dependence of stress incidence.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is a disease with restricted cognitive memory function and intellectual skills, which occurs after surgery with and without anesthesia. The limiting cognitive ability leads to a lack of quality of life for a lot of patients. The POCD strongly depends on patient's age and the surgical operation type. In aged adults the incidence of POCD after one week following surgery is 25,8%. Risk factors for the development of a POCD is beside age less education and a reduced cognitive reserve. However, the anesthesia procedure plays a pivotal role as well and regarding the current knowledge it is still uncertain which technique matches the lowest risk. Elevated stress level accompanied with regional anesthesia procedures are accused to cause POCD in elderly patients. This fact leads to the question if a general anesthesia technique has a lower stress level and consequently leads to a reduced risk for a POCD development. Likewise the investigators address this hypothesis and analyze cognitive function following both anesthesia techniques separately in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 50-85 years of age both gender.

Exclusion Criteria:

* Patients under 50 years of age or older than 85 years of age.
* Preexisting neurological, neuropsychological deficits or diseases, e.g. cerebral insult or epilepsy.
* Preexisting neurological, neuropsychological medication, preexisting neuromuscular diseases.
* Alcohol- and drug abuse. Postoperative complications, pain and time shifts within the test protocol.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients recruted at the University Hospital Erlangen prior surgery. Anesthesia procedure eigther in regional or general manner.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Function | 5 Days
  Using different tests addressing a various quality of neurocognitive function (attention, memory, perceptual and processing speed, alertness and executive function) participants score test appropriate values. Comparing test values separately allows to distinguish between prior - and post - operative status. Moreover it allows to discriminate achieved test results between both groups and calculate statistical differences. Favorable test results lead to a potential better neurocognitive function outcome and enable to assess neurocognitive function in the light of operation consequence.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Dept. Anaesthesiology, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Wagner S, Breitkopf M, Ahrens E, Ma H, Kuester O, Thomas C, von Arnim CAF, Walther A. Cognitive function in older patients and their stress challenge using different anesthesia regimes: a single center observational study. BMC Anesthesiol. 2023 Jan 6;23(1):6. doi: 10.1186/s12871-022-01960-7. PMID 36609226